CLINICAL TRIAL: NCT04983212
Title: Peri-implantitis in HIV-positive Patients With Different Dental Prosthesis
Acronym: PERIHIV
Status: Completed | Type: Observational
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Luca Casula, MD, Msc, Università Vita-Salute San Raffaele
Other Study IDs: 10/INT/2020
Record Dates: First submitted 2021-07-08; First posted 2021-07-30 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Peri-Implantitis
Keywords: peri-implantitis; HIV-positive; Mucositis
MeSH Terms: conditions — Peri-Implantitis; HIV Seropositivity; Mucositis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: periodontal control — patient were called and visited in the dentistry department and gingival sulcus were gentle probed to assess gingiva and peri-implant tissues status

SUMMARY:
Dental implants are widely used in human immunodeficiency virus (HIV)-positive patients, but the interaction between immune status and success of implant therapy, especially in such patients, is not clear.

This study aimed to assess the prevalence of peri-implantitis in HIV-positive patients and to evaluate the presence of a possible correlation between the immunological profile and serological values of the same HIV-positive patients, of peri-implantitis, and of possible differences between all-on-4 and single crown/bridge prostheses in terms of peri-implant disease and the variables analyzed.

This cross sectional study included 85 adult HIV-positive patients (394 implants) with at least one dental implant loaded for more than a year who were followed for at least one year. The patients were divided into patients with all-on-4 prosthesis and those with single crowns/bridges to assess the differences between the two types of prostheses in the inflammatory state, in the presence of mucositis and peri-implantitis, and in the variables analyzed. The following clinical parameters were assessed: full-mouth plaque score (FMPS), full-mouth bleeding score (FMBS), probing pocket depth (PPD) in six sites per implant and tooth (deepest value for each implant and tooth was registered), PI and BoP measured as presence/absence at six sites per implant and tooth, presence of suppuration, mobility (measured by manual palpation) and number of lost teeth.

DETAILED DESCRIPTION:
2.1 Study design This cross-sectional mono-centric observational study assessed the prevalence of peri-implant disease in HIV-positive patients and was performed in accordance with the Helsinki Declaration of Human Studies. All procedures were approved by the Ethics Committee of Vita-Salute San Raffaele University (on 15/7/2020 with number of protocol "PERIHIV"-EC Reg. N. 10/INT/2020) in Milan, Italy. This study has been reported according to the STrengthening the Reporting of OBservational studies in Epidemiology (STROBE) guidelines and checklist.

2.2 Patient sample Each patient was informed about all pertinent aspects of the study by the investigator (LC), and an appropriate informed consent was obtained prior to the start of the study. The study included 85 adult patients between 46.56 and 55.6 years (median 51.32 years) with at least one dental implant and a total of 394 dental implants with a mean follow-up of 3 years (range from 2 years to 5 years). Demographic, clinical, and laboratory information of the patients was collected and implant were positioned in the same Hospital in which patients are in treating with antiretroviral therapy for the HIV-infection (Ville Turro Dental Clinic of Vita-Salute San Raffaele University in Milan).

2.3 Inclusion and exclusion criteria All patients (>18 years old) who had undergone prosthetic rehabilitation using one or more dental implants, with at least 1 year of follow-up after loading, and who had returned for a maintenance appointment at the Ville Turro Dental Clinic of Vita-Salute San Raffaele University in Milan. All patients were undergoing antiretroviral therapy (ART) at the same hospital. Patients who discontinued antiretroviral therapy and patients not undergoing therapy, subjects with uncontrolled systemic diseases (diabetes [HbA1c>7]) or under treatment with any medications that may have an effect on bone turnover and mucosal healing (steroids, bisphosphonate therapy ) were excluded. Pregnancy or breastfeeding women were also excluded. All patients were included in a maintenance oral hygiene program (every 4 months) and who discontinued the oral maintenance (more than 1 appointment) were excluded from the study.

2.4 surgery procedure All implants were placed by two skilled implant surgeons; most of the implants (328) were 3,8 mm diameter (83.2%), 46 were 3,3 mm (11.7%) and 20 were 4,5 mm (5.1%). Implants were placed at level or slightly below the bone crest (1 mm) and in all cases the complete bone healing was reached (at least 3 months) before implant loading. Bone healing was assessed after at least 3 months of undisturbed healing, with periapical radiographs and if confirmed, final impression was taken. For implant-supported single crown and bridge, after final impression, definitive cemented single crown or bridge were achieved. Only in cases of not adequate prosthetic space, with not sufficient abutment retention for cemented prostheses, screw-retained prosthetic rehabilitations were made. Regarding the full arch rehabilitations, the all-on-four protocol described by Malò were followed in all cases. In addition the bone was leveled before implant placement using a rongeur and with the aid of the carbide burs in order to form a flat bone plane in which place the implant. This allows the elimination of the bone spicules, fractured bone and damaged buccal bone and the creation of a flatbed in which was easy to insert the implants and achieve the prosthetic rehabilitation. Two implants were placed in the posterior sectors (tilted) and two in the anterior sector (straight) after the bone leveling.

2.4 Clinical evaluation Data pertaining probing pocket depth (PPD), bleeding on probing (BoP) and plaque index (PI) around the implants and teeth of HIV-positive patients included in the study were collected by probing implant and dental sulcus with a calibrated dental probe (0,25 N)(Hawe Click-Probe®, KerrHawe SA, Switzerland) by one skilled operator (L.C.). The following clinical parameters were assessed: full-mouth plaque score (FMPS), full-mouth bleeding score (FMBS), probing pocket depth (PPD) in six sites per implant and tooth (deepest value for each implant and tooth was registered), PI and BoP measured as presence/absence at six sites per implant and tooth, presence of suppuration, mobility (measured by manual palpation) and number of lost teeth. Demographic data and implant site characteristics were checked in a specific case report form. For each HIV-positive patients, the following information was reported: age, gender, smoking habit (number of cigarettes), number of dental implants, health condition (i.e. diabetes presence), history of periodontitis and frequency of maintenance (number of maintenance appointments in 1 year). Data relating to the immunological and systemic profile of the patients (HIVRNA load, CD4+ level, CD8+ level, hemoglobin level, platelet count) were collected through the database of the hospital.

For each implant, the following data were collected: diameter, location, time in function, type of prosthesis (crown/bridge or all-on-4). The patients were divided into two groups, according to the type of prosthesis inserted after implant placement, to assess the differences between the two types of prostheses in the inflammatory state, and therefore, in the presence of mucositis and peri-implantitis as well as in the variables analyzed.

2.5 Radiologic examination and assessment of bone level When an implant showed BoP with or without suppuration and/or PPD ≥ 3 mm after gentle probing, a periapical radiograph was taken using the long-cone paralleling technique and using Rinn rings for the periapical images. The position of the marginal bone was measured manually on ultra speed radiographic film (Ultra speed, Kodak, USA) using a dental caliper (0 to 10 mm) and with the aid of 4.5X magnification (EyeMag Pro F, Zeiss). The distance to the marginal bone was measured at the mesial and distal aspects of the implants to the adjacent bone. The implant platform was used as reference for the measurements. Two vertical lines were drawn parallel to the vertical line crossing the centre of the implant. The largest value was recorded. Assessments were performed by one investigator (PC).

2.6 Case definitions for peri-implant conditions The criteria described in 2017 in Periodontology World Workshop by Renvert (2018) were used for peri-implant disease diagnosis: Peri-implant mucositis was diagnoses in presence of visual inspection demonstrating the presence of peri-implant signs of inflammation, presence of profuse bleeding and/or suppuration on probing; an increase in probing depths compared to baseline and absence of bone loss in relation to the baseline.

Peri-implantitis was diagnoses in presence of bleeding on probing and/or suppuration, increasing probing pocket depths as compared to measurements obtained at placement of the supra-structure and progressive bone loss in relation to the radiographic bone level assessment at 1 year following the delivery of the implant-supported prosthetics reconstruction. In the absence of initial radiographs and probing depths, radiographic evidence of bone levels ≥ 3 mm apical of the most coronal portion of the intra-osseous part of the implant and/or probing depths ≥6 mm in conjunction with profuse bleeding were used for the diagnosis. Gentle probing.

2.7 Case definitions for history of periodontitis The criteria described in 2017 in Periodontology World Workshop by Tonetti (2018) were used for history of periodontitis diagnosis: Presence of periodontitis was detected as clinical attachment loss (CAL) with reference to the cemento-enamel junction (CEJ) not ascribed to non-periodontal causes.

1. Interdental CAL detectable at ≥ 2 non-adjacent teeth
2. Buccal or oral CAL ≥3 mm with pocketing >3 mm detectable at ≥2 teeth CAL was assessed with the periodontal probing or with direct visualization to detect the CEJ. Moreover to confirm the CAL periapical radiographs and/or rx OPT were used.

ELIGIBILITY:
Inclusion Criteria:

* patients (>18 years old) who had undergone prosthetic rehabilitation using one or more dental implants, with at least 1 year of follow-up after loading, and
* patients who had returned for a maintenance appointment at the Ville Turro Dental Clinic of Vita-Salute San Raffaele University in Milan
* patients under antiretroviral therapy (ART) at the same hospital.

Exclusion Criteria:

* Patients who discontinued antiretroviral therapy
* patients not undergoing therapy
* patients with uncontrolled systemic diseases (diabetes [HbA1c>7])
* patients under treatment with any medications that may have an effect on bone turnover and mucosal healing (steroids, bisphosphonate therapy )
* Pregnancy or breastfeeding women
* patients who discontinued the oral maintenance (more than 1 appointment)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with detected HIV infection and under retroviral therapy (HAART) that had positioned at least 1 dental implant with at least one year follow-up
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
prevalence of peri-implantitis | 01/01/2015 - 01/01/2020
  peri-implantitis is characterized by inflammation of the peri-implant mucosa associated with a progressive loss of supporting bone

CONTACTS AND LOCATIONS:
Locations (1):
- Ville Turro, San Raffaele Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No